CLINICAL TRIAL: NCT01942590
Title: A Clinical Investigation of the Safety and Efficacy of Clenbuterol on Motor Function in Individuals With Late-onset Pompe Disease and Receiving Enzyme Replacement Therapy
Brief Title: Safety and Efficacy of Clenbuterol in Individuals With Late-onset Pompe Disease and Receiving Enzyme Replacement Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dwight Koeberl, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Dwight Koeberl, M.D., Ph.D., Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00043680; R01FD004364 (FDA)
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Pompe Disease
Keywords: Pompe disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Clenbuterol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clenbuterol (Experimental): Initially, 40 mcg each morning for one week. Then, increase to 40 mcg BID for the next 5 weeks. If tolerated, will increase to 80 mcg in the morning and 40 mcg in the evening for one week. Then, last dose increase will be 80 mcg BID until week 52.
  Interventions: Drug: Clenbuterol
- Placebo Comparator (Placebo Comparator): Initially, one capsule each morning for one week. Then, increase to one capsule BID for the next 5 weeks. If tolerated, will increase to two capsules in the morning and one capsule in the evening for one week. Then, last dose increase will be two capsules BID until week 52.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clenbuterol
  Other Names: Spiropent
  Arms: Clenbuterol
Drug: Placebo
  Other Names: Capsule
  Arms: Placebo Comparator

SUMMARY:
Funding Source- FDA OOPD

The purpose of this study is to investigate the safety and efficacy of clenbuterol on motor function in individuals with late-onset Pompe disease (LOPD) who are treated with enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
This is a 52 week Phase I/II double-blind, randomized, placebo-controlled study of adjunctive clenbuterol in LOPD (Table 2, Section 6). All subjects will be evaluated at Week 0 and Week 6 to establish a baseline for motor function testing. At Week 6, subjects will be randomized 3:2 to clenbuterol or placebo, and evaluated for safety and efficacy during the Week 12 and 18 visits. The Investigational Drug Service will maintain double-blinding by providing either the study drug or placebo (over-encapsulated tablets) directly to subjects. The drug (or placebo) will be initiated at the Week 6 visit in a staged manner (first once daily and later BID), and the dose will be increased at the Week 12 visit in a similarly staged manner to minimize AEs and related attrition. All subjects will return for a final visit after a total of 52 weeks in the study.

In terms of standard of care, the subject will have two clinical visits (charged to the subject and/or the subject's insurance company), one at the initiation of the study drug (baseline) and one at the study completion (52 weeks). Study drug will be attempted to be initiated during the "off week", approximately one week following a dose of ERT, and ERT will continue throughout the duration of the study. Thereafter, study visits will be during the "off week". The 6, 12, and 18 week visits will be research visits (not charged to the subject and/or the subject's insurance company) in order to determine subject's overall health status and measure early signs of motor improvement. The initial dose of clenbuterol will be 40 mcg per oral each morning for one week, followed by 40 mcg BID for the next 5 weeks until the week 12 visit. If the 40 mcg BID per oral is well tolerated, the dose will be increased to 80 mcg each morning/40 mcg each evening for one week, followed by 80 mcg BID for the next 5 weeks until the Week 18 visit. If 80 mcg BID is tolerated at Week 18, the subject will continue on that dose until Week 52.

Compliance will be discussed at the Week 6, Week 12, and Week 18 visits. The subject will have phone visits during Week 1, 7, 13, 36, and 52, and compliance will be discussed then. We will call subjects daily during the first week following initiation of study drug (Week 7) and dosage escalation (Week 13) to support subjects through the early adverse effects of tachyphylaxis that may lead to premature termination. An interim call will occur during Week 36 to monitor compliance. Subjects who admit non-compliance, missing >6 doses of the study drug, will be considered non-compliant and withdrawn from the study. Subjects will be called during Week 1 and Week 52, 3 days following the muscle biopsy. All phone calls will review AEs (Table).

The efficacy of clenbuterol treatment during ERT in patients with LOPD will be evaluated with muscle and pulmonary function testing as the primary endpoints. A secondary endpoint, the urinary Glc4 biomarker, will be monitored when the subjects are evaluated at baseline, week 18 and week 52. The impact of enhanced CI-MPR-mediated uptake of GAA will be analyzed by comparing the muscle function, pulmonary function, and biochemical correction of muscle in subjects with LOPD treated with ERT, both prior to and during simultaneous β2 agonist therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Pompe disease by blood acid alpha-glucosidase assay and acid alpha-glucosidase gene sequencing,
2. Age: 18+ years at enrollment,
3. Receiving ERT at standard dose (20 mg/kg every 2 weeks) for at least 52 weeks,
4. Subjects are capable of giving written consent.

Exclusion Criteria:

1. Continuous invasive ventilation (via tracheostomy or endotracheal tube)
2. Clinically relevant illness within two weeks of enrollment including fever > 38.2 C, vomiting more than once in 24 hours, seizure, or other symptom deemed contraindicative to new therapy.
3. Chronic heart disease (Myocardial infarction, arrythmia, cardiomyopathy)
4. Tachycardia
5. History of seizure disorder
6. Hyperthyroidism
7. Pheochromocytoma
8. Pregnancy
9. History of diabetes
10. History of hypersensitivity to beta 2-agonist drugs such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline, salmeterol (Serevent),
11. Patients on a non-standard schedule for ERT; for example, weekly infusions as opposed to infusions every two weeks.
12. Treatment for asthma in the previous 12 months.
13. The use of the following concommitant meds is prohibited during the study:

    * diuretics (water pill);
    * digoxin (digitalis, Lanoxin);
    * beta-blockers such as atenolol (Tenormin), metoprolol (Lopressor), and propranolol (Inderal);
    * tricyclic antidepressants such as amitriptyline (Elavil, Etrafon), doxepin (Sinequan), imipramine (Janimine, Tofranil), and nortriptyline (Pamelor);
    * Monoamine oxidase inhibitors such as isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam), or tranylcypromine (Parnate); or
    * other bronchodilators such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline (Brethine, Bricanyl), salmeterol (Serevent), isoetherine (Bronkometer), metaproterenol (Alupent, Metaprel), or isoproterenol (Isuprel Mistometer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09-02 (Actual); Study Completion 2016-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight D Koeberl, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Kamalakkannan G, Petrilli CM, George I, LaManca J, McLaughlin BT, Shane E, Mancini DM, Maybaum S. Clenbuterol increases lean muscle mass but not endurance in patients with chronic heart failure. J Heart Lung Transplant. 2008 Apr;27(4):457-61. doi: 10.1016/j.healun.2008.01.013. PMID 18374884
- [Background] Koeberl DD, Luo X, Sun B, McVie-Wylie A, Dai J, Li S, Banugaria SG, Chen YT, Bali DS. Enhanced efficacy of enzyme replacement therapy in Pompe disease through mannose-6-phosphate receptor expression in skeletal muscle. Mol Genet Metab. 2011 Jun;103(2):107-12. doi: 10.1016/j.ymgme.2011.02.006. Epub 2011 Feb 13. PMID 21397538
- [Background] Koeberl DD, Li S, Dai J, Thurberg BL, Bali D, Kishnani PS. beta2 Agonists enhance the efficacy of simultaneous enzyme replacement therapy in murine Pompe disease. Mol Genet Metab. 2012 Feb;105(2):221-7. doi: 10.1016/j.ymgme.2011.11.005. Epub 2011 Nov 11. PMID 22154081
- [Derived] Koeberl DD, Case LE, Smith EC, Walters C, Han SO, Li Y, Chen W, Hornik CP, Huffman KM, Kraus WE, Thurberg BL, Corcoran DL, Bali D, Bursac N, Kishnani PS. Correction of Biochemical Abnormalities and Improved Muscle Function in a Phase I/II Clinical Trial of Clenbuterol in Pompe Disease. Mol Ther. 2018 Sep 5;26(9):2304-2314. doi: 10.1016/j.ymthe.2018.06.023. Epub 2018 Jul 5. PMID 30025991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 participants signed consent; 13 participants were randomized.
Groups:
- Clenbuterol: Initially, 40 mcg each morning for one week. Then, increase to 40 mcg BID for the next 5 weeks. If tolerated, will increase to 80 mcg in the morning and 40 mcg in the evening for one week. Then, last dose increase will be 80 mcg BID until week 52.
  Clenbuterol
- Placebo Comparator: Initially, one capsule (placebo) each morning for one week. Then, increase to one capsule BID for the next 5 weeks. If tolerated, will increase to two capsules in the morning and one capsule in the evening for one week. Then, last dose increase to two capsules until week 52.
  Placebo
Period: Overall Study
Arm/Group | Clenbuterol | Placebo Comparator
Started | 8 | 5
Completed | 7 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clenbuterol: Initially, one capsule (40 mcg) each morning for one week. Then, increase to 40 mcg BID for the next 5 weeks. If tolerated, will increase to 80 mcg in the morning and 40 mcg in the evening for one week. Then, last dose increase will be 80 mcg BID until week 52.
  Clenbuterol
- Total: Total of all reporting groups
Arm/Group | Clenbuterol | Placebo Comparator | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 65] | 32 [19 to 62] | 51 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Creatine Kinase (CK) Reflecting Worsening of Muscle Involvement
Description: Worsening muscle involvement, as defined by >3x increase in CK from baseline that is >2x the upper limit of normal
Time Frame: Any point up to week 52
Measure: Number; unit: participants
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 8 | 5
participants | 1 | 0

2. Primary Outcome: Number of Participants With a Change in Aspartate Aminotransferase (AST), Alanine Transaminase (ALT), and Bilirubin Representing Liver Toxicity
Description: Liver toxicity, as defined by a >3x increase in AST or ALT from the respective baseline values and/or an increase in direct, indirect or total bilirubin of >3x the upper limit of normal
Time Frame: Any point up to week 52
Measure: Number; unit: participants
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 8 | 5
participants | 0 | 0

3. Secondary Outcome: Change in 6 Minute Walk Test
Description: Assess exercise tolerance in study patients; test administered by physical therapist. Subjects were asked to walk for 6 minutes, unassisted. The distance walked was recorded in meters.
Time Frame: Baseline, week 18
Population: Participants who completed 6 minute walk test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 4
meters | 18.09 (24.85) | 6.878 (76.02)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.0512, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.434, t-test, 1 sided

4. Secondary Outcome: Change in 6 Minute Walk Test
Description: as for outcome 3
Time Frame: Baseline, week 52
Population: Participants who completed 6 minute walk test
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 6 | 4
meters | 16.42 (24.61) | -18.13 (40.9)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.0816, t-test, 1 sided — Paired t test comparing each subject's performance at Week 52 to Baseline
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.3318, t-test, 1 sided — Paired t test comparing each subject's performance at Week 52 to Baseline

5. Secondary Outcome: Change in Forced Vital Capacity (FVC) in Pulmonary Function Testing
Description: Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.
Time Frame: Baseline, Week 18
Population: participants who completed FVC testing
Measure: Mean (Standard Deviation); unit: change in FVC measured as % expected
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 8 | 4
change in FVC measured as % expected | 1.575 (5.14) | 2.825 (11.78)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.2074, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.332, t-test, 1 sided

6. Secondary Outcome: Change in Forced Vital Capacity (FVC) in Pulmonary Function Testing
Description: Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.
Time Frame: Baseline, Week 52
Population: participants who completed FVC testing
Measure: Mean (Standard Deviation); unit: change in FVC measured as % expected
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 4
change in FVC measured as % expected | -5.738 (20.04) | 7.775 (11.98)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.233, t-test, 1 sided — Paired t test comparing each subject's performance at Week 52 to Baseline
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.142, t-test, 1 sided — Paired t test comparing each subject's performance at Week 52 to Baseline

7. Secondary Outcome: Change in Urinary Glc4 Biomarker
Description: The Glc4 biomarker is measured in urine and correlates with muscle glycogen content. It is a noninvasive measurement that serves as a biomarker for Pompe disease.
Time Frame: Baseline, Week 18
Measure: Mean (Standard Deviation); unit: mmol/mol CN
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 3 | 4
mmol/mol CN | -1.733 (0.6028) | 0.0667 (0.666)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.019, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.366, t-test, 1 sided

8. Secondary Outcome: Change in Urinary Glc4 Biomarker
Time Frame: Baseline, Week 52
Population: participants who completed urinary Glc4 biomarker collection
Measure: Mean (Standard Deviation); unit: mmol/mol CN
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 6 | 3
mmol/mol CN | -1.1 (1.857) | -1.667 (2.401)
Statistical Analysis 1: Comparison: Clenbuterol; Test type: Other; p = 0.161, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo Comparator; Test type: Other; p = 0.43, t-test, 1 sided

9. Secondary Outcome: GSGC (Gait, Stairs, Gowers, Arising From a Chair.)
Description: The GSGC is a criterion referenced assessment designed to measure functional status and change in gross motor function over time and, in particular, to measure clinically relevant change. Consists of 4 components: Gait, Climbing Stairs, Gower's Manuever, Arising From a Chair. Lowest score 4 = normal muscle function, highest score 27 = unable to perform motor function tests.
Time Frame: Baseline, Week 18, and Week 52
Population: participants who completed GSGC testing
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 4
units on a scale
  Baseline | 17 (4.69) | 7.5 (5.07)
  Week 18 | 15.14 (5.61) | 6.5 (3.7)
  Week 52: number analyzed (Participants) | 6 | 4
  Week 52 | 13.8 (5.6) | 6.5 (3)
Statistical Analysis 1: Comparison: Clenbuterol; Baseline, week 18; Test type: Other; p = 0.01, t-test, 1 sided
Statistical Analysis 2: Comparison: Clenbuterol; Baseline, week 52; Test type: Other; p = 0.004, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo Comparator; Baseline, week 18; Test type: Other; p = 0.154, t-test, 1 sided
Statistical Analysis 4: Comparison: Placebo Comparator; Baseline, Week 52; Test type: Other; p = 0.211, t-test, 1 sided

10. Secondary Outcome: Quick Motor Function Test (QMFT)
Description: The QMFT is a criterion referenced assessment designed to measure functional status and change in gross motor function over time and, in particular, to measure clinically relevant change. Consists of 16 motor function tests. Lowest score 0 = unable to perform motor function tests, highest score 64 = normal muscle function.
Time Frame: Baseline, Week 18, and Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 5 | 4
units on a scale
  Baseline | 35 (16.4) | 53.75 (13.7)
  Week 18 | 40.6 (17.97) | 54.75 (14.08)
  Week 52 | 46.5 (15.1) | 56.25 (14.2)
Statistical Analysis 1: Comparison: Clenbuterol; Baseline, Week 18; Test type: Other; p = 0.006, t-test, 1 sided
Statistical Analysis 2: Comparison: Clenbuterol; Baseline, Week 52; Test type: Other; p = 0.007, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo Comparator; Baseline, Week 18; Test type: Other; p = 0.297, t-test, 1 sided
Statistical Analysis 4: Comparison: Placebo Comparator; Baseline, Week 52; Test type: Other; p = 0.196, t-test, 1 sided

11. Secondary Outcome: Late-Life Function and Disability Instrument (LLFDI)
Description: The Late-Life Function & Disability Instrument (Late-Life FDI) is an evaluative outcome instrument for community-dwelling older adults. Highest score 240 = normal function and no disability, lowest score 0 = low levels of frequency of participating in life tasks.
Time Frame: Baseline, Week 18, Week 52
Population: Participants who completed LLFDI at the visit. Data was not collected from any participants in the placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 4 | 0
units on a scale
  Baseline | 103.75 (26.81) |
  Week 18: number analyzed (Participants) | 3 | 0
  Week 18 | 106.7 (39.3) |
  Week 52 | 112.5 (27.4) |
Statistical Analysis 1: Comparison: Clenbuterol; Baseline Week 18; Test type: Other; p = 0.3639, t-test, 1 sided
Statistical Analysis 2: Comparison: Clenbuterol; Baseline, Week 52; Test type: Other; p = 0.0371, t-test, 1 sided

12. Secondary Outcome: Predicted Maximum Inspiration Pressure (MIP)
Description: MIP is a measurement of inspiratory muscle weakness, including weakness of the diaphragm. MIP is decreased in Pompe disease and reflects weakness of respiratory muscles.
Time Frame: Baseline, Week 18, and Week 52
Population: Participants who completed the MIP testing
Measure: Mean (Standard Deviation); unit: percentage of MIP
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 4
percentage of MIP
  Baseline | 56.3 (34.64) | 96.8 (17.23)
  Week 18 | 47.4 (20.19) | 83.8 (15.13)
  Week 52: number analyzed (Participants) | 6 | 4
  Week 52 | 68.5 (26.86) | 104.6 (13.9)
Statistical Analysis 1: Comparison: Clenbuterol; Baseline, Week 18; Test type: Other; p = 0.268, t-test, 1 sided
Statistical Analysis 2: Comparison: Clenbuterol; Baseline, Week 52; Test type: Other; p = 0.0036, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo Comparator; Baseline, Week 18; Test type: Other; p = 0.286, t-test, 1 sided
Statistical Analysis 4: Comparison: Placebo Comparator; Baseline, Week 52; Test type: Other; p = 0.279, t-test, 1 sided

13. Secondary Outcome: Maximum Expiratory Pressure (MEP)
Description: MEP reflects the strength of the abdominal muscles and other expiratory muscles.
Time Frame: Baseline, Week 18, and Week 52
Population: Participants who completed the MEP testing
Measure: Mean (Standard Deviation); unit: percentage of MEP
Arm/Group | Clenbuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 4
percentage of MEP
  Baseline | 40.4 (17.5) | 62.8 (14.5)
  Week 18: number analyzed (Participants) | 7 | 3
  Week 18 | 40 (16.8) | 83.3 (30.4)
  Week 52: number analyzed (Participants) | 6 | 4
  Week 52 | 53.9 (7.8) | 49.2 (11.6)
Statistical Analysis 1: Comparison: Clenbuterol; Baseline, Week 18; Test type: Other; p = 0.479, t-test, 1 sided
Statistical Analysis 2: Comparison: Clenbuterol; Baseline, Week 52; Test type: Other; p = 0.059, t-test, 1 sided
Statistical Analysis 3: Comparison: Placebo Comparator; Baseline, Week 18; Test type: Other; p = 0.152, t-test, 1 sided
Statistical Analysis 4: Comparison: Placebo Comparator; Baseline, Week 52; Test type: Other; p = 0.118, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: baseline to 52 week
Arm/Group | Clenbuterol | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/5
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clenbuterol (N=8) | Placebo Comparator (N=5)
fall (Musculoskeletal and connective tissue disorders) | 1 | 0 — Dislocated artificial hip
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clenbuterol (N=8) | Placebo Comparator (N=5)
anxiety (General disorders) | 2 | 1
decreased appetite (General disorders) | 2 | 0
Elevated creatine kinase (>3x baseline) (Musculoskeletal and connective tissue disorders) | 1 | 0
GI upset (Gastrointestinal disorders) | 2 | 0
weight gain (General disorders) | 2 | 0
increased urination frequency (Renal and urinary disorders) | 3 | 0
Insomnia (General disorders) | 5 | 2
Muscle spasma (Musculoskeletal and connective tissue disorders) | 4 | 1
Palpitations (Cardiac disorders) | 2 | 1
Tremors (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes